CLINICAL TRIAL: NCT06109870
Title: Prevención en Sus Manos: Feasibility of a Novel Community-Based Strategy to Improve Access to Cervical Cancer Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0529; NCI-2023-09607 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: HPV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRECEDE-PROCEED (Experimental): To identify predisposing, enabling, and reinforcing factors that could influence women's decision to participate in self-sample HPV testing and diagnostic follow-up.
  Interventions: Behavioral: PRECEDE-PROCEED

INTERVENTIONS:
Behavioral: PRECEDE-PROCEED — delivered self-sampling (CHWSS) to increase screening participation.

SUMMARY:
Cervical cancer is a disease that is preventable through vaccination against the virus that causes it, human papillomavirus (HPV), and through screening and treatment of cervical disease before it becomes cancet.

DETAILED DESCRIPTION:
Primary Objectives:

The overall purpose of this protocol is to evaluate the feasibility and acceptability of CHW-delivered selfsample HPV testing (CHW-SS) to increase cervical cancer screening among women in RGV and other low- resource communities in Texas.

The specific aims of this protocol are to:

Specific Aim 1: Determine the feasibility of CHW-SS in the RGV and other low-resource communities in Texas (i.e., reach, screening uptake, notification of test results).

Specific Aim 2: Assess the acceptability and experiences of CHW-SS among under screened persons in rural, persistent poverty communities in the RGV and other low-resource communities in Texas.

Secondary Objectives:

Exploratory Aim 3: Assess attendance for clinical follow-up among individuals who participate in CHW-SS and test positive for HR-HPV.

Exploratory Aim 4: Evaluate contextual fit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Currently resident in RGV or other low-resource community in Texas
* Stated willingness to comply with all study procedures
* Females; Age ≥25 years
* Have no history of hysterectomy with removal of the cervix
* Have no history of cervical cancer or high-grade dysplasia
* Have not had a Pap test in the past 3.5 years or Pap/HPV co-test in the past 5.5 years.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Unable to communicate in English or Spanish
* Lack valid telephone contact information
* Report being currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Montealegre, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Texas at Austin, Austin, Texas
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fallah PN, Bowman P, Tran C, Chen V, Pippin M, Varon ML, Baker E, Milan J, Parker SL, Lezama-Sierra J, Munsell MF, Desravines N, Lavie I, Batman S, Montealegre J, Schmeler KM, Williams-Brown MY, Salcedo MP. Implementation of Human Papillomavirus Self-Collection and Barriers to Follow-Up Among Unhoused Individuals in Texas: The EMPOWER Study. Obstet Gynecol. 2025 Nov 1;146(5):710-717. doi: 10.1097/AOG.0000000000006003. Epub 2025 Jul 17. PMID 40674748
- See also: M D Anderson Cancer Center — http://www.mdanderson.org